CLINICAL TRIAL: NCT00508781
Title: Multiphoton Laser Scanning Microscopy in Cutaneous Optical Pathology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Other Study IDs: 9100206857
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2007-07-30 (Estimated); Status verified 2002-11

CONDITIONS: Optical Biopsy; Cutaneous Pathology; Dermatopathology

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Multiphoton laser image in cutaneous pathology

SUMMARY:
We use multiphoton laser scanning microscopy to observe cutaneous anatomy and pathology. The study aims to compare surgical specimen by conventional pathology slice with the image by non-invasive multiphoton laser scanning microscopy.

DETAILED DESCRIPTION:
For skin diseases, the most convincing method for diagnosis to date is surgical biopsy. However, a skin biopsy is an invasive procedure which carries the risk of tissue damage, wound infection and scar formation. To solve the inconvenience from surgical biopsy, multiphoton laser scanning microscopy is a developing, non-invasive method for observing the cutaneous anatomy and pathology. Multiphoton laser scanning microscopy is good in tissue penetration and resolution with less tissue damage. The study aims to compare surgical specimen by conventional pathology slice with the image by non-invasive multiphoton laser scanning microscopy. A good correlation in multiphoton image may serve as optical biopsy for cutaneous pathology and spare the invasive procedure of skin biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving cosmetic surgeries such as removal of moles

Exclusion Criteria:

* No special exclusion criteria

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2002-11; Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shiou-Hwa Jee, MD PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan